CLINICAL TRIAL: NCT05895019
Title: Effects of Propofol on Brain Function in Patients With Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Other Study IDs: ywn20220901
Record Dates: First submitted 2023-05-02; First posted 2023-06-08 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: PD - Parkinson's Disease
Keywords: Propofol; Electroencephalography; Cerebral autoregulation
MeSH Terms: conditions — Parkinson Disease | interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Parkinson's disease: Patients with Parkinson's disease
  Interventions: Drug: Propofol
- Non-Parkinson's patients: Non-Parkinson's patients
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol was administered using TCI pump induction with a starting target effect concentration of 1.0ug/ml. The target concentration was increased by 0.2-0.5ug/ml if the patient did not reach unconsciousness after 1 min of stabilization of the target concentration. The propofol concentration recorded at this time was the target concentration the patient was induced to unconsciousness. The state of consciousness was tested every 60 s by the investigator, and clinical trial data were collected for 5 min; after that, clinical trial data were recorded before and after induction of anesthesia at 5 min after induction of anesthesia, at intubation and skin dissection, and 1, 3, and 5 min after intubation and skin dissection, respectively.

SUMMARY:
Propofol is a short-acting general anesthetic drug commonly used in clinical practice, with rapid clinical onset of action, amnesic, anxiolytic, antiepileptic, and muscle relaxant effects. The lack of natural antioxidants in patients with Parkinson's disease and propofol's ability to protect the brain by inhibiting oxidative stress, its pharmacokinetic and pharmacodynamic properties make propofol a suitable anesthetic drug for functional stereotactic surgery in patients with Parkinson's disease. However, changes in brain functional status during propofol anesthesia in Parkinson's patients are unknown. There is a lack of data from extensive clinical studies to support the need for propofol dosing during induction of anesthesia compared with non-Parkinson patients. This study is a prospective cohort study designed to compare the differences in propofol dosing requirements during induction of propofol anesthesia in patients with PD versus non-PD and to monitor the characteristics of altered brain functional status such as EEG and cerebral blood flow autoregulation capacity in PD versus non-PD patients during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

PD group:

1. age 18-80 years, ASA class I-III, proposed bilateral DBS surgery;
2. primary PD, or hereditary PD, various genotypes of PD, responding well to compounded levodopa;
3. informed consent obtained;

Non-PD group:

1. age 18-80 years, ASA class I-III, proposed non-neurosurgical non-cardiac surgery;
2. no previous clearly diagnosed neurological disease or neurological dysfunction;
3. informed consent obtained.

Exclusion Criteria:

1. Obstructive sleep apnea;
2. BMI > 30kg/m2;
3. Estimated difficult airway;
4. Patients with prior allergy to anesthetic drugs;
5. Serious dysfunction of important organs (i.e. heart failure, renal or liver dysfunction);
6. Patients with craniocerebral trauma or craniocerebral operation history resulting in incomplete skull or brain parenchyma defect;
7. Patients with alcohol or drug addiction.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: PD group: (1) age 18-80 years, ASA class I-III, proposed bilateral DBS surgery; (2) primary PD, or hereditary PD, various genotypes of PD, responding well to compounded levodopa; (3) informed consent obtained; Non-PD group: (1) age 18-80 years, ASA class I-III, proposed non-neurosurgical non-cardiac surgery; (2) no previous clearly diagnosed neurological disease or neurological dysfunction; (3) informed consent obtained.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Propofol Dose | During the trial(up to 30 minutes for each subject)
  Differences in propofol dose required during induction of propofol anesthesia in Parkinson's disease versus non-Parkinson's disease patients

SECONDARY OUTCOMES:
Feature extraction of EEG Signals | During the trial(up to 3 hours for each subject)
  To compare the correlation between OAA/S sedation scores and EEG and its quantitative indexes
Feature Extraction of EEG Signals | During the trial(up to 3 days for each subject)
  To compare the EEG power in delta、theta、alpha and beta band
Cerebral Autoregulation | During the trial(up to 3hours for each subject)
  The mean velocity of the middle cerebral artery，transient hyperemic response ratio
Patient Satisfaction with Sedation | During the trial(up to 3 days for each subject)
  to assess patient satisfaction with sedation and the occurrence of adverse events during sedation on a four-level scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided